CLINICAL TRIAL: NCT02482389
Title: A Phase II Study of Preoperative Boost Radiotherapy in Patients With Breast With Biomarker Analysis
Brief Title: Study of Preoperative Boost Radiotherapy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of enrollment
Sponsor: Duke University (Other)
Collaborators: Gateway for Cancer Research (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00063936
Record Dates: First submitted 2015-06-22; First posted 2015-06-26 (Estimated); Results first posted 2022-03-23 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-03

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm 7 Gray (Gy) fraction of radiotherapy (Experimental): All subjects will receive a single 7 Gy fraction of radiotherapy to the intact tumor prior to surgery.
  Interventions: Radiation: Single fraction of 7 Gy

INTERVENTIONS:
Radiation: Single fraction of 7 Gy — All subjects will receive a single 7 Gy fraction of radiotherapy to the intact tumor prior to surgery.

SUMMARY:
This protocol seeks to utilize a novel method of tumor bed boost delivery and to better understand breast cancer radiation response through the analysis of pre-and post-radiation breast tumor samples.

DETAILED DESCRIPTION:
The study team proposes in this trial to build on the favorable results of the intraoperative boost trials but using a preoperative delivery approach. The PI has demonstrated the feasibility of the preoperative approach and successfully completed a Phase I dose-finding partial breast trial. The preoperative approach has several advantages: 1) expensive intra-operative equipment is unnecessary, 2) a small intact breast tumor results in significantly less uninvolved breast tissue receiving high radiation doses which likely decreases toxicity; 3) more accurate targeting of the high-risk areas of subclinical disease surrounding the tumor is possible, 4) smaller treatment volumes are amenable to dose escalation which can further accelerate treatment and improve accessibility for subjects, and 5) the pre-operative approach provides a novel opportunity to study breast cancer radiation response.

Radiotherapy to the intact tumor is a relatively rare event in breast cancer irradiation, particularly in the setting of early stage breast cancer. Tumor and normal tissue radiation response remain relatively poorly understood. Markers capable of predicting radiation response are rare indeed. Therefore, paired pre- and post-radiation tissue will be examined for FAS gene expression and compared among the breast cancer subtypes. FAS is the name of a gene ( not an acronym) that is known to play a critical role in the induction of programmed cell death and is an established prognostic marker in breast cancer. Previous study team findings that FAS induction appears to be breast cancer subtype-specific has not been previously observed and provides a possible explanation for the differential rates of tumor response observed clinically in distinct breast tumor subtypes. The study team's preclinical work with FAS suggests a potential role as a radiation response biomarker. The study goal is to validate those findings in this large cohort of diverse breast cancer subjects. However, because preoperative delivery of the boost to the intact tumor is unique, this study will include a secondary cosmetic outcome that includes predefined stopping boundaries for early indications of suboptimal cosmetic outcomes with this novel approach

ELIGIBILITY:
Inclusion Criteria:

1. Women with a biopsy proven diagnosis of ductal carcinoma in situ or invasive carcinoma of the breast. Biopsy tissue (either slides or block) from outside institutions will be reviewed to confirm diagnosis.
2. Breast preservation candidates (no prior breast or nodal radiotherapy, no imaging evidence of multicentric disease preventing resection through a single incision, no pregnant women, and no comorbid conditions precluding surgery)
3. cTis-T3 cancer judged to benefit (by treating radiation oncologist) from a tumor bed boost
4. Women of child-bearing potential must consent to use adequate contraception during the course of the study: (1) surgical sterilization (such as a tubal ligation or hysterectomy), (2) approved hormonal contraceptives (such as birth control pills, patches, implants or injections), (3) barrier methods (such as a condom or diaphragm) used with a spermicide, or (4) an intrauterine device (IUD). Contraceptive measures such as Plan B (TM), sold for emergency use after unprotected sex, are not acceptable methods for routine use.
5. White blood cell (WBC) > 3000, Hgb > 10, platelets >100000 within 30 days of consent
6. Eligible for contrasted magnetic resonance imaging( MRI) on initial evaluation with glomerular filtration rate (GFR) ≥ 60 ml/min. A diagnostic MRI ordered within 60 days of diagnosis will be considered an acceptable alternative and will not be repeated.
7. Outside breast imaging will be reviewed at Duke to confirm that findings are consistent with trial eligibility

Exclusion Criteria:

1. Breast implant in the breast to be treated (contralateral breast implant is acceptable)
2. Medical conditions that may increase risk for poor cosmetic outcome (i.e. Lupus, rheumatoid arthritis, scleroderma)
3. Subjects unable to receive study treatment planning secondary to body habitus or inability to lie flat on the stomach for at least 1 hour
4. Positive serum pregnancy test
5. Insufficient breast imaging to judge clinical stage
6. Subjects without placement of a biopsy clip at the diagnostic procedure who are unwilling to undergo clip placement.
7. Subjects in whom treatment planning constraints cannot be met

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 3 (Actual)
Dates: Start 2015-09-08 (Actual); Primary Completion 2021-06-25 (Actual); Study Completion 2021-06-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Blitzblau, MD PhD, Principal Investigator — Duke Health
Locations (1):
- Duke Cancer Center, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Single Arm 7 Gray (Gy) Fraction of Radiotherapy
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Single Arm 7 Gray (Gy) Fraction of Radiotherapy
Number analyzed (Participants) | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.67 (3.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Cosmesis evaluation [Mean (Standard Deviation); unit: units on a scale] — Cosmesis score is calculated using the NRG Oncology cosmesis scale which reports physical appearance from 1 (excellent) to 4 (poor), with a lower score representing a better outcome.
  units on a scale | 1 (0)

OUTCOME MEASURES:

1. Primary Outcome: Change in Cosmesis Evaluations Using the NRG Oncology Cosmesis Scale
Description: Change from baseline rates of cosmesis at 3 years post-treatment as measured by the NRG Oncology cosmesis scale. The scale is scored from 1 (excellent) to 4 (poor) with a lower number representing better physical appearance.
Time Frame: baseline to 3 years post radiation therapy
Measure: Number (95% Confidence Interval); unit: score on a scale
Arm/Group | Single Arm 7 Gray (Gy) Fraction of Radiotherapy
Number analyzed (Participants) | 3
score on a scale | 0 [0 to 0]

2. Secondary Outcome: Change Circulating Cell Free DNA to Identify Potential Radiation Response Biomarkers
Description: Blood collected pre and post treatment will be used to explore the biologic response to radiotherapy by comparing changes in circulating cell-free DNA expression pre and post-radiotherapy:
Time Frame: 5 years
Population: Data not collected.
Arm/Group | Single Arm 7 Gray (Gy) Fraction of Radiotherapy
Number analyzed (Participants) | 0

3. Secondary Outcome: Quality of Life as Measured by Functional Assessment of Cancer Therapy - Breast (FACT-B) Questionnaire
Description: Patient-reported Quality of Life as measured by the Functional Assessment of Cancer Therapy - Breast (FACT-B) at 3 years post-treatment. The FACT-B includes 35 items scored on a Likert-type scale from 0 (not at all) to 4 (very much) with a total scale range of 0-140 and a lower total score indicating a better outcome. Only the total scale score is reported; subscales scores are not reported.
Time Frame: 3 years
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Single Arm 7 Gray (Gy) Fraction of Radiotherapy
Number analyzed (Participants) | 3
score on a scale | 11.7 (7.5)

4. Secondary Outcome: Composite Review of Local Control
Description: Document local control in the treated breast relative to historical controls with annual clinical exam and imaging studies. Local control is defined as the time from start of treatment to date of local recurrence estimated using the Kaplan-Meier method.
Time Frame: 5-10 years
Population: Data will not be collected and reported as the study was terminated prematurely due to poor accrual.
Arm/Group | Single Arm 7 Gray (Gy) Fraction of Radiotherapy
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | Single Arm 7 Gray (Gy) Fraction of Radiotherapy
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 3/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm 7 Gray (Gy) Fraction of Radiotherapy (N=3)
Breast pain (Reproductive system and breast disorders) | 2 (4)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 2 (3)
Fibrosis deep connective tissue (Musculoskeletal and connective tissue disorders) | 2 (4)
Seroma (Injury, poisoning and procedural complications) | 1 (1)
Other (Reproductive system and breast disorders) | 1 (1) — Palpable cording on the underside of the right upper arm
Bruising (Injury, poisoning and procedural complications) | 2 (2)
Other (Injury, poisoning and procedural complications) | 1 (1) — open scar, no sign of infection

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-20): https://cdn.clinicaltrials.gov/large-docs/89/NCT02482389/Prot_SAP_000.pdf